CLINICAL TRIAL: NCT04962607
Title: Effectiveness of Premixed Bioactive Bioceramic MTA (Neo-Putty®) Versus Formocresol as Dressing Agents in Pulpotomized Primary Molars
Brief Title: Effectiveness of Premixed Bioactive Bioceramic MTA (Neo-Putty®) in Pulpotomies Primary Teeth
Status: Active, not recruiting | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: 0994-20-HMO
Record Dates: First submitted 2021-06-28; First posted 2021-07-15 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Pulpotomies on Primary Molars

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Study Group: 1. Asymptomatic primary molars with deep carious lesions scheduled for regular treatment.
  2. Exposure of a vital pulp due to caries.
  3. No clinical or radiographic evidence of pulp degeneration, such as spontaneous pain, excessive bleeding from the root canal, internal root resorption, inter-radicular and/or periapical bone destruction, swelling, or sinus tract.
  4. The possibility of proper restoration of the teeth.
  Interventions: Other: Neo-Putty® as dressing agents in pulpotomized primary molars
- control group: 1. Asymptomatic primary molars with deep carious lesions scheduled for regular treatment.
  2. Exposure of a vital pulp due to caries.
  3. No clinical or radiographic evidence of pulp degeneration, such as spontaneous pain, excessive bleeding from the root canal, internal root resorption, inter-radicular and/or periapical bone destruction, swelling, or sinus tract.
  4. The possibility of proper restoration of the teeth.
  Interventions: Other: Neo-Putty® as dressing agents in pulpotomized primary molars

INTERVENTIONS:
Other: Neo-Putty® as dressing agents in pulpotomized primary molars — Following removal of the coronal pulp with a round bur and hemostasis, the pulp stumps in the study group will be covered with Neo-Putty ® according to the manufacturer's instructions. Neo-Putty will be placed in the prepared cavity, and then covered with Vitrebond® and with a reinforced Zinc Oxide-Eugenol (IRM, Bayer-Leverkussen, Germany).
  In the control group, a cotton pellet moistened with full-strength FC will be placed for 5 minutes on the amputated pulp, after reaching hemostasis. The pulp stumps will be then covered by IRM

SUMMARY:
The objective of this prospective randomized clinical trial is to assess clinically and radiographically, the effect of NeoPutty as a pulp medicament following coronal pulp amputation in human primary molars with carious pulp exposure in comparison to Formocresol (FC).

ELIGIBILITY:
Inclusion Criteria:

* primary teeth which requires pulpotomy.

Exclusion Criteria:

* not healthy patients,
* teeth which requires pulpectomy.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy children attending the Pediatric Dentistry Clinic of the Hebrew University-Hadassah School of Dental Medicine in Jerusalem
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Success rate of the primary molar pulpotomy | One year

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No